CLINICAL TRIAL: NCT02340884
Title: A Pilot Randomized Controlled Trial of the Promoting Resilience in Stress Management (PRISM) Intervention for Adolescents and Young Adults With Cancer
Brief Title: A Pilot RCT of the PRISM Intervention for AYAs With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Abby Rosenberg, Associate Professor, Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SC-N114
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Acute Lymphoblastic Leukemia; Lymphoma; Sarcoma; Acute Myelogenous Leukemia; Brain Tumors; Germ Cell Tumor
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Sarcoma; Leukemia, Myeloid, Acute; Brain Neoplasms; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRISM (Experimental): Promoting Resilience In Stress Management Intervention (skills-based intervention designed to teach stress-management, goal-setting, cognitive reframing, and meaning-making skills)
  Interventions: Behavioral: Promoting Resilience In Stress Management (PRISM)
- Control (No Intervention): Standard psychosocial supportive care

INTERVENTIONS:
Behavioral: Promoting Resilience In Stress Management (PRISM) — The brief format of the PRISM intervention involves 4, 50-minute, one-on-one sessions approximately 2 weeks apart, plus a 5th parent-inclusive session 2-4 weeks following session #4. These are complimented with age-specific handouts describing the skills and opportunities to practice them, as well as weekly (text- or email based) check-ins from study staff and in-person "booster" sessions once monthly. Specifically, the intervention incorporates four primary skills: 1) stress management/mindfulness; 2) goal-setting; 3) cognitive restructuring; and, 4) meaning-making/benefit finding.
  Arms: PRISM

SUMMARY:
Study Title: A Pilot Randomized Controlled Trial of the Promoting Resilience in Stress Management (PRISM) Intervention for Adolescents and Young Adults with Cancer

Study Population and Sample Size: Two cohorts of Adolescent and Young Adult (AYA) patients with diagnosis of new or recurrent cancer between 1 and 10 weeks prior to enrollment: those ages 13-17 (N=50); (2) those ages 18-25 (N=50).

Study Design: Pilot randomized controlled trial (RCT).

Primary Objective: To test the efficacy of the "Promoting Resilience in Stress Management" (PRISM) among Adolescents and Young Adults with cancer.

Primary Outcome: Change in patient-reported resilience (based on score of standardized Connor-Davidson Resilience Scale) at 6 months.

Secondary Outcomes:

1. Patient-reported resilience at 2, 4, and 12 months
2. Patient-reported self-efficacy, benefit-finding, psychological distress, quality of life, and health-behaviors at 6 and 12 months.
3. Qualitative assessment of patient-reported goals at 6 and 12 months
4. Development of a cohort of AYA cancer survivors for assessment of long-term psychosocial outcomes

Study Duration: 3 years

DETAILED DESCRIPTION:
The experience of serious illness among adolescents and young adults (AYAs) is unique because they face distinctive developmental challenges, transitions, and choices related to education, employment, identity, relationships and family. Age-specific interventions are needed to promote positive resources and outcomes. Resilience, for example, is a construct describing an individual's capacity to maintain psychological and/or physical well-being in the face of stress, and is a good candidate to buffer the negative effects of stress. While few studies have described positive outcomes in AYA patients with chronic disease, and fewer still have suggested mechanisms to promote resilience, evidence suggests promoting "resilience-resources" (e.g., stress-management and goal setting skills, meaning-making and positive-reframing of negative experiences), as a means to manage stress may be valuable.

We have previously described models and factors of resilience among AYAs with cancer as well as parents of children with cancer, and demonstrated that self-perceptions of resilience are strongly associated with outcomes. Through iterative pilot testing, we have successfully developed a novel, patient-centered resilience-based intervention, the "Promoting Resilience in Stress Management" (PRISM) intervention.

The overall goal of the PRISM intervention is to improve AYA self-perceived resilience, thereby reducing AYA distress, improving quality of life, and minimizing risky health behaviors. The brief format involves 4, 50-minute, one-on-one sessions approximately 2 weeks apart, plus a 5th, optional, family-inclusive session 2-4 weeks following session #4. These are complimented with age-specific handouts describing the skills and opportunities to practice them, as well as monthly "booster" sessions. Specifically, the intervention incorporates four primary skills: 1) stress management/mindfulness; 2) goal-setting; 3) cognitive restructuring; and, 4) meaning-making/benefit finding.

Enrolled patients will be between 13 and 25 years-old with at least a 2 week history of new or recurrent malignancy. They will be randomized to receive the PRISM intervention or standard psychosocial supportive care. Patients in both groups will be invited to complete quantitative surveys at the time of enrollment and then 2-, 4-, 6-, and 12-months later. Participants will be compensated for their time.

The primary outcome of the study is self-perceived resilience, as measured by the Connor-Davidson Resilience Score, at 6-months post-enrollment. Secondary outcomes will assess resilience scores at 4, 6, and 12 months, as well as self-efficacy, anxiety, depression, benefit-finding, quality of life, goal-setting skills, and health behaviors at 6 and 12 months.

The study is anticipated to accrue a total of 100 patients over 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-25 years

   1. Patient aged 13-17 years: has signed informed assent and their parent/legal guardian has signed informed consent for study participation.
   2. Patient aged 18-25 years: has signed informed consent for study participation.
2. Diagnosis of malignancy treated with chemotherapy and/or radiation therapy at Seattle Childrens Hospital (SCH)

   1. New diagnosis of malignancy within 1-10 weeks of enrollment
   2. New diagnosis of recurrent disease (after initial remission) within 1-10 weeks of enrollment
3. Ability to speak and read English language
4. Cognitively able to participate in interactive interviews

Exclusion Criteria:

1. Patient refusal to participate (any age), or parental refusal to participate for patients less than 18 years of age
2. Cognitively or physically unable to participate in interactive interview
3. Unable to speak and read English language
4. Patient without chemotherapy and/or radiation therapy as part of cancer treatment (e.g., surgical resection only patients are not-eligible).

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Resilience | 6 months

SECONDARY OUTCOMES:
Patient-Reported self-efficacy | 6 months
Patient-Reported benefit-finding | 6 months
Patient-Reported goal-setting skills | 6 months
Patient-Reported quality of life | 6 months
Patient-Reported health behaviors | 6 months
Patient-reported anxiety & depression | 6 months

OTHER OUTCOMES:
Patient-reported resilience | 4- and 6- months

CONTACTS AND LOCATIONS:
Overall Officials: Abby R Rosenberg, MD, MS, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Rosenberg AR, Zhou C, Bradford MC, Salsman JM, Sexton K, O'Daffer A, Yi-Frazier JP. Assessment of the Promoting Resilience in Stress Management Intervention for Adolescent and Young Adult Survivors of Cancer at 2 Years: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2136039. doi: 10.1001/jamanetworkopen.2021.36039. PMID 34817581
- [Derived] Steineck A, Barton KS, Bradford MC, Yi-Frazier JP, Rosenberg AR. Tincture of Time: The Evolution of Goals in Adolescents and Young Adults with Cancer. J Adolesc Young Adult Oncol. 2021 Dec;10(6):703-710. doi: 10.1089/jayao.2020.0223. Epub 2021 May 6. PMID 33960833
- [Derived] Lau N, Bradford MC, Steineck A, Scott S, Bona K, Yi-Frazier JP, McCauley E, Rosenberg AR. Examining key sociodemographic characteristics of adolescents and young adults with cancer: A post hoc analysis of the Promoting Resilience in Stress Management randomized clinical trial. Palliat Med. 2020 Mar;34(3):336-348. doi: 10.1177/0269216319886215. Epub 2019 Nov 4. PMID 31680625
- [Derived] Lau N, Bradford MC, Steineck A, Junkins CC, Yi-Frazier JP, McCauley E, Rosenberg AR. Exploratory analysis of treatment response trajectories in the PRISM trial: Models of psychosocial care. Psychooncology. 2019 Jul;28(7):1470-1476. doi: 10.1002/pon.5098. Epub 2019 May 14. PMID 31037789